CLINICAL TRIAL: NCT00344292
Title: SNPs and Extent of Atherosclerosis (SEA) Study
Brief Title: Understanding the Genetic and Hereditary Basis of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1333; U01HL080443-01A1 (NIH); R01 HL080443-01A1
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-03

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Polymorphism, Genetic; Coronary Artery Disease; Coronary Arteriosclerosis; Polymorphism, Single Nucleotide; SNPs
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Atherosclerosis is a condition that occurs when fatty deposits build up along the inner walls of arteries. New strategies are needed to prevent and treat atherosclerosis. The purpose of this study is to analyze the DNA of participants in two ongoing studies to identify genetic variations responsible for the development of atherosclerosis.

DETAILED DESCRIPTION:
Atherosclerosis is a condition in which deposits of fat, cholesterol, and other substances build up along the inner walls of arteries; these deposits are known as plaque. As plaque builds up, it increases the risk of blood clots, heart attack, and stroke. Research has shown that the risk of developing atherosclerosis can be influenced by heredity. However, researchers have been unable to identify the specific genes associated with this risk. Single nucleotide polymorphisms (SNPs) are small genetic variations that can occur within an individual's DNA. In this study, researchers will analyze the DNA of many individuals for differences in SNP patterns. The goal of the study is to determine which SNP patterns are associated with the development of atherosclerosis. The data from this study may lead to new strategies for early identification of high risk individuals who may benefit from aggressive treatment to prevent the development of atherosclerosis.

This study will not recruit any new participants. DNA will be collected and analyzed from participants in two existing studies-the Pathobiological Determinants of Atherosclerosis in Youth (PDAY) study and the Multi-Ethnic Study of Atherosclerosis (MESA). DNA from the PDAY participants will be obtained from liver samples gathered during an autopsy following the participants' deaths; DNA from the MESA participants will be obtained from blood collected during routine study visits. There will be no additional study visits for participants, and all DNA samples and study information will be kept confidential. Genetic testing will be performed to determine the association between SNPs and subclinical atherosclerosis, which is a form of the condition prior to the onset of symptoms. The study will evaluate specific variations in SNPs and subclinical disease among different ethnic groups, which may help to explain why certain ethnic groups have higher rates of atherosclerosis. The study will also examine the association between SNPs and other indicators of subclinical and clinical atherosclerosis, including the thickness of arteries, heart calcium levels, and blood pressure levels.

ELIGIBILITY:
Inclusion Criteria:

* Participant in PDAY or MESA

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject enrolled in the Pathobiologic Determinants of Atherosclerosis in Youth (PDAY) study
Sampling Method: Non-Probability Sample
Enrollment: 2763 (Actual)
Dates: Start 2006-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To estimate the association between common single nucleotide polymorphisms (SNPs) in the human genome and extent of subclinical atherosclerosis among subjects in the Pathobiological Determinants of Atherosclerosis in Youth (PDAY) cohort (N=2,876). | Entire project period.
To estimate the association between potential atherosclerosis SNPs identified in the PDAY cohort and extent of subclinical atherosclerosis among subjects in the Multi-Ethnic Study of Atherosclerosis (MESA) cohort (N=6,577). | Entire project period
To define the haplotypic structure of the genome in the regions of SNPs that are associated with atherosclerosis in PDAY and MESA and to perform additional genotyping necessary for haplotype association studies using both the PDAY and MESA cohorts. | Entire project period.
To disseminate the identity, location, primer sets and allele frequency of the atherosclerosis associated SNPs in PDAY, and those confirmed in MESA, in order to facilitate additional replication and functional studies of the most promising SNPs. | Entire project period.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Herrington, MD, MHS, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Cedars-Sinai Health System, Los Angeles, California
  - Louisiana State University, New Orleans, Louisiana
  - The University of Texas, Houston, Texas
  - University of Washington, Seattle, Washington